CLINICAL TRIAL: NCT05564169
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of Masitinib as add-on Therapy in Patients With Mild Alzheimer's Disease, Treated With Standard of Care
Brief Title: Masitinib in Patients With Mild Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB21004
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Mast Cells; Microglia; Tyrosine kinase inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — masitinib; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Parallel group (1:1), Multicenter, Comparative study over 24 weeks with a 24-week extension period (all patients can enter the extension phase until week 48).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerized central randomization system using an external provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib (4.5) & SOC (Experimental): Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment. Dose up-titration is subjected to a safety control. Masitinib will be administered as an add-on to cholinesterase inhibitor and/or memantine standard of care (SOC).
  Interventions: Drug: Masitinib (4.5); Drug: Standard of care
- Placebo & SOC (Placebo Comparator): Participants receive a matched dose placebo, given orally twice daily. Placebo will be administered as an add-on to cholinesterase inhibitor and/or memantine standard of care (SOC).
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Placebo — treatment per os
  Other Names: Placebo Oral Tablet
  Arms: Placebo & SOC
Drug: Masitinib (4.5) — Masitinib (titration to 4.5 mg/kg/day)
  Other Names: AB1010
  Arms: Masitinib (4.5) & SOC
Drug: Standard of care — Cholinesterase inhibitors (donepezil, rivastigmine or galantamine) and/or memantine

SUMMARY:
Masitinib is an orally administered tyrosine kinase inhibitor that targets activated cells of the neuroimmune system (mast cells and microglia). Study AB21004 will evaluate masitinib as an adjunct to cholinesterase inhibitor and/or memantine in patients with mild-to-moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Masitinib is an oral tyrosine kinase inhibitor that has demonstrated neuroprotective action in neurodegenerative diseases via inhibition of mast cell and microglia/macrophage activity, and which is capable of accumulating within the central nervous system (CNS) at a therapeutically relevant concentration. There is a growing body of evidence implicating mast cells and microglia (types of innate immune cells that are present in the CNS), with the pathophysiology of Alzheimer's disease.

Masitinib has been shown to restore normal spatial learning performance and promote recovery of synaptic markers in a mouse model of Alzheimer's disease, with its synapto-protective action being directly linked to mast cell inhibition. The potential benefit of masitinib in the treatment of patients with mild to moderate Alzheimer's disease has been previously demonstrated in a phase 2 study (AB04024; NCT00976118) and a positive phase 2B/3 study (AB09004; NCT01872598) that showed masitinib (4.5 mg/kg/day) was associated with a statistically significant slowing of cognitive deterioration.

The objective of study AB21004 is to confirm treatment effect with masitinib as an adjunct to cholinesterase inhibitor and/or memantine in patients with mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Main inclusion criteria include:

1. Patient with clinical diagnosis of Alzheimer's disease based on criteria defined by IWG (International Working Group on Alzheimer's disease) at screening visit.
2. Patients with ADCS-ADL score at screening visit and baseline visit < 73
3. Patient with MMSE ≥ 21 and ≤ 25 at screening visit and baseline visit.
4. Patient with Alzheimer's Disease biomarker profile at screening visit:

   * A positive amyloid PET scan
   * Alternatively, positive a-beta AND p-tau results OR an abnormal p-tau/a-beta ratio in CSF analysis. Before randomization, the results will be verified centrally.
5. If patients are treated with cholinesterase inhibitors (donepezil, rivastigmine or galantamine), and/or memantine. They should have been at stable dose for a minimum of 6 months at baseline visit, with no changes foreseen in therapy throughout the trial.
6. If receiving a supplement for cognition (eg, gingko biloba, omega-3 polyunsaturated fatty acid, vitamin E, curcumin, souvenaid) patients must have been taking it at stable dose for at least 4 months prior to screening visit.
7. Patients with a caregiver who, at screening and baseline visits, agrees to accompany the participant to all trial visits, supervise compliance with procedures, provide detailed information, has sufficient contact (≥1 hour/day for ≥3 days/week or as deemed sufficient by the Investigator), can read, understand, and speak the designated language, and is cognitively capable of fulfilling trial requirements.

Main exclusion criteria include:

Related to disease

1. Patients with any other cause of dementia shown by MRI findings and neurological examination
2. Systemic conditions known to cause dementia, e.g., hypothyroidism, untreated vitamin B12 or folic acid deficiency, niacin deficiency, neurosyphilis, HIV infection at screening visit.
3. Patients with substance-induced dementia, Alzheimer's disease with delirium, severe delusions (e.g., NPI delusion score ≥ 4), psychosis or antipsychotic use, or a history of significant psychiatric disorders at the screening visit.
4. Patients with a significant unexplained improvement or decline in overall status on ADAS-Cog and ADCS-ADL at screening and baseline compared to previous assessments, and those whose scores are not in line with their medical history.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in iADRS score at week 24 | 24 weeks
  The iADRS is a linear combination of its two components: the ADAS-Cog11 and the ADCS-iADL. The iADRS is calculated as follows: iADRS = ADCS-iADL + (70 - ADAS-Cog11).
  Lower scores on the iADRS indicate greater impairment; iADRS scores range from 0 to 129.

SECONDARY OUTCOMES:
Absolute change from baseline in Mini-Mental State Examination (MMSE) at week 24 | 24 weeks
  Mini-Mental State Examination (MMSE) (scores from 0 to 30, with lower scores indicating poorer cognitive performance)
Absolute change from baseline in ADAS-Cog11 score at week 24 | 24 weeks
  The global score, which is the sum of the 11 items, ranges from 0 to 70, with higher scores indicating greater cognitive impairment.
Absolute change from baseline in ADCS-ADL score | 48 weeks
  Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory scale (ADCS-ADL) (scores from 0 to 78, with lower scores indicating worse function)
Clinical Responder rate | 24 weeks
  Clinical response defined as decrease from baseline at week 24 in ADAS-cog of ≥4, without deterioration in ADCS-ADL (ADCS-ADL change ≥ 0 between baseline and timepoint) or worsening in the CIBIC-plus scale (response CIBIC in 1-3] or no change [CIBIC in 4]).
CIBIC-plus | 24 weeks
  Clinician's Interview-Based Impression of Change plus Caregiver Input (CIBIC-plus), a seven-point categorical rating scale ranging from 1 (marked improved) to 7 (markedly worse) compared with baseline.
Absolute change from baseline in CDR | 24 weeks
  Clinical Dementia Rating (CDR), scores from 0 to 18, with higher scores indicating worse dementia
Time to severe dementia (MMSE<10) | 24 weeks
  Mini-Mental State Examination (MMSE) (scores from 0 to 30, with lower scores indicating poorer cognitive performance)
Absolute change from baseline in ADAS-Cog11 score at week 48 | 48 weeks
  The global score, which is the sum of the 11 items, ranges from 0 to 70, with higher scores indicating greater cognitive impairment.
Absolute change from baseline in ADCS-ADL score at week 24 | 24 weeks
  Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory scale (ADCS-ADL) (scores from 0 to 78, with lower scores indicating worse function)
Absolute change from baseline in Neuropsychiatric Inventory (NPI) at week 24 | 24 weeks
  Total NPI-12 score ranges from 0 to 144 (higher = more severe symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, MD, PhD, Principal Investigator — Hôpital Universitaire Pitié-Salpêtrière, Paris, France
Locations (9):
- Institut de la mémoire et Maladie d'Alzheimer, Hôpitaux Universitaires Pitié-Salpêtrière, Paris, France
- Spain (8):
  - Hospital Universitario Nuestra Señora del Perpetuo Socorro de Albacete (Hospital Universitario Nuestra Señora del Perpétuo Socorro), Albacete
  - Ace Alzheimer Center Barcelona (Fundació ACE), Barcelona
  - Hospital Policlínico de Gipuzkoa, Donostia / San Sebastian
  - Virgen de las Nieves University Hospital (Hospital Universitario Virgen de las Nieves), Granada
  - La Paz University Hospital (Hospital Universitario La Paz), Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Navarra, Pamplona
  - Complejo Asistencial de Zamora. Hospital Provincial de Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piette F, Belmin J, Vincent H, Schmidt N, Pariel S, Verny M, Marquis C, Mely J, Hugonot-Diener L, Kinet JP, Dubreuil P, Moussy A, Hermine O. Masitinib as an adjunct therapy for mild-to-moderate Alzheimer's disease: a randomised, placebo-controlled phase 2 trial. Alzheimers Res Ther. 2011 Apr 19;3(2):16. doi: 10.1186/alzrt75. PMID 21504563
- [Background] Dubois B, Lopez-Arrieta J, Lipschitz S, Doskas T, Spiru L, Moroz S, Venger O, Vermersch P, Moussy A, Mansfield CD, Hermine O, Tsolaki M; AB09004 Study Group Investigators. Masitinib for mild-to-moderate Alzheimer's disease: results from a randomized, placebo-controlled, phase 3, clinical trial. Alzheimers Res Ther. 2023 Feb 28;15(1):39. doi: 10.1186/s13195-023-01169-x. PMID 36849969
- [Background] Li T, Martin E, Abada YS, Boucher C, Ces A, Youssef I, Fenaux G, Forand Y, Legrand A, Nachiket N, Dhenain M, Hermine O, Dubreuil P, Delarasse C, Delatour B. Effects of Chronic Masitinib Treatment in APPswe/PSEN1dE9 Transgenic Mice Modeling Alzheimer's Disease. J Alzheimers Dis. 2020;76(4):1339-1345. doi: 10.3233/JAD-200466. PMID 32623401